CLINICAL TRIAL: NCT07214597
Title: NICU Utilization of Remote Voice Technology to Improve mateRnal Experience (NURTURE): A Randomized Controlled Trial
Brief Title: NICU Utilization of Remote Voice Technology to Improve mateRnal Experience (NURTURE)
Acronym: NURTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Osmundson, Associate Professor in Obstetrics and Gynecology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 251461; 4R42MH135602-02 (NIH)
Record Dates: First submitted 2025-09-04; First posted 2025-10-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Depression (PPD); Self-Efficacy; Parental Anxiety; Engagement, Patient; Usability; Length of Stay
Keywords: Neonatal Intensive Care Unit; NICU; Postpartum Depression (PPD); VoiceLove app; NURTURE; VoiceLove
MeSH Terms: conditions — Depression, Postpartum; Patient Participation

STUDY DESIGN:
Intervention Model Description: Infant/mother dyads will be randomized in a 1:1 ratio stratified by infant gestational age at delivery (<28 vs ≥28 weeks) and depression/anxiety diagnosis of the mother (measured by baseline EPDS ≥13). Gestational age is strongly associated with infant length of NICU stay. To reduce the risk of selection bias, we will use allocation concealment employing a computer-generated, permuted-block randomization scheme with varying block size. The block size and randomization list will only be known to the biostatistician creating the randomization list and will not be shared with investigators or any other study personnel. This list will be directly uploaded into REDCap's randomization module. Treatment assignment will be known by study participants, research personnel, and medical team given the unblinded nature of the intervention. Randomization procedure details, including stratification and block sizes, will be reported in trial publications. Randomization assignments are accessible 27/4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm (Experimental): Participants in this arm will be randomized to receive access to the VoiceLove app in addition to standard of care.
  Interventions: Device: VoiceLove mobile phone application
- Control Arm (No Intervention): Participants in this arm will be randomized to standard of care only and will not have access to the VoiceLove app.

INTERVENTIONS:
Device: VoiceLove mobile phone application — Access to VoiceLove app to facilitate secure, real-time communication between family members and NICU patients.
  Other Names: VoiceLove app
  Arms: Intervention Arm

SUMMARY:
The study's objective is to conduct a Phase II randomized controlled trial examining the preliminary efficacy of the VoiceLove app compared to usual care on maternal postpartum depression in mothers with infants admitted to the Neonatal Intensive Care Unit (NICU). Primary aim: Assess the effects of VoiceLove on maternal postpartum depression, measured by the Edinburgh Postnatal Depression Scale (EPDS). The estimates from this study will be used for a future definitive Phase III trial. Secondary aim: Assess feasibility, acceptability, and patterns of communication and engagement among mothers, partners, and NICU clinicians during the NICU hospitalization, measured through app usage metrics, satisfaction surveys, and qualitative interviews. Additionally, we will evaluate effects of infant length of stay.

DETAILED DESCRIPTION:
This study is a randomized control trial that will test VoiceLove, a secure mobile app designed to help families communicate with their infants in the Neonatal Intensive Care Unit (NICU).

Postpartum depression (PPD) is a major depressive disorder and is one of the most frequent childbirth complications. Mother-infant separation during the initial postpartum period, such as infant admission to the neonatal intensive care unit (NICU), impacts mother-infant bonding and increases PPD risk, which is 40% higher in mothers with children admitted to the NICU. The impact of PPD is substantial: reported poor quality of life, high-risk behaviors such as substance abuse or self-harm, and long-term impairments in child cognitive and emotional development. PPD impact on child development has potential to be magnified in the already vulnerable preterm infant population. Care in the NICU is, by design, focused on the health of the infant and ill-equipped to address parental mental health. High stress and burnout among NICU staff combined with limited resources for development of psychosocial programs targeting the parents of NICU patients underscore the need for simple, low-cost, and easily implemented interventions aimed at improving parental connectedness and reducing postpartum mental health disorders.

Lack of parental connectedness to their neonate during a NICU stay and low social support are two of the most powerful risk factors for developing PPD. Risk of PPD is decreased when parents have more contact, either physical or verbal, with their infant and a higher perceived social support system. When physical contact is not possible, voice contact may help foster feelings of connectedness to both the infant in the NICU, and to the parents' social circle. The medical team is another critical source of support poised to increase parental mental health. Mothers of infants in the NICU report increased depressive symptoms when their perception of nurse support is low, while increased communication between parents and the medical team improves parental well-being. Increased social support from loved ones and the medical care team is well positioned to significantly reduce PPD severity in parents of NICU infants. Thus, facilitation of communication between parents and healthcare providers, as well as between their friends and family, presents a low-cost, low effort means to dramatically impact parental mental health and well-being during a NICU admission.

VoiceLove Inc has developed a novel HIPAA-compliant mobile application that offers programmatic support and curated digital content (e.g., lullabies, music, environmental sounds) for infant-family interactions and enables expanded family engagement in hospital settings. VoiceLove mobile app circumvents barriers to communication through an electronic venue for direct patient-family-clinician interaction. Specifically for clinicians, VoiceLove is a safe and time-efficient tool for direct communication with absent family members, allowing more time for direct patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Infant:

   1. Admitted to the neonatal intensive care unit (NICU)
   2. Born at VUMC
   3. Index admission (NOT a re-admission)
   4. Born between 23+0 and 31+6 weeks
   5. Expected to survive at least 2 weeks
   6. Singleton gestation
2. Mother:

   1. Age ≥ 18 years old
   2. English speaking
   3. Mother is the biological mother of the infant admitted to the NICU
   4. Postpartum day 4 or less
3. Partner (NOTE: Partner enrollment is not required)

   1. Mother agrees to partner's participation
   2. Designated by mother as support person with infant access

Exclusion Criteria

1. Infant

   a. Re-admission to NICU
2. Mother

   1. No access to an Android or iOS smartphone
   2. Unwilling to download the VoiceLove NICU app to their personal smartphone and unwilling to accept the terms and conditions of the VoiceLove app
   3. No personal email address
   4. Incarcerated at time of delivery or postpartum
   5. Inability to obtain informed consent

   i. Patient's clinician refuses enrollment of the patient ii. Patient is either mentally (acute psychosis) or physically (intubated or critically ill in the ICU) unable to provide informed consent f. Unable to approach the patient (staffing, patient unavailable) g. Mother is not the intended parent (plans adoption, is a surrogate, will not have custody of the infant)
3. Partner (NOTE: Partner enrollment is not required)

   1. Age < 18 years old
   2. Not English speaking
   3. Inability to obtain informed consent
   4. No access to an Android or iOS smartphone that is different from the mother's smartphone
   5. No access to an email address that is different from the mother's email address
   6. Unwilling to download the VoiceLove NICU app to their personal smartphone and unwilling to accept the terms and conditions of the VoiceLove app

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient Engagement with the VoiceLove App | 2-weeks post randomization.
  To assess the feasibility of using the VoiceLove app, we will measure how much patients in the intervention group engage with the app using metrics such as average app use per day at 2-weeks post randomization.
Edinburgh Postnatal Depression Score (EPDS) at 2-weeks post randomization. | 2-weeks post randomization.
  The EPDS is a 10-question assessment of postpartum depression measured continuously on a scale of 1 to 30, whereas a higher score is a higher indication of postpartum depression.

SECONDARY OUTCOMES:
EPDS Score at 6-weeks post randomization | 6-weeks post randomization.
  The EPDS is a 10-question assessment of postpartum depression measured continuously on a scale of 1 to 30, whereas a higher score is a higher indication of postpartum depression.
Prevalence of high risk for postpartum depression (EPDS score ≥ 13) at 2- and 6-weeks. | 2- and 6-weeks post randomization
  Edinburgh Postnatal Depression Score (EPDS) ≥ 13. The EPDS is a 10-question assessment of postpartum depression measured continuously on a scale of 1 to 30, whereas a higher score is a higher indication of postpartum depression.
PROMIS Informational Support at 2- and 6-weeks post randomization | 2- and 6-weeks post randomization
  Patient-Reported Outcomes Measurement Information System (PROMIS). According to HealthMeasures, the following describes the PROMIS Informational Support: "Quality of social support refers to functional aspects of supportive relationships, i.e., interpersonal relationships that serve particular functions. This includes the interactive process by which emotional, instrumental or informational support is obtained from one's social network. It also includes companionship, feeling cared for and valued as a person, communication with others, and feelings of belonging and trust. Measures of social support generally seek information about a person's perception of the availability or adequacy of resources provided by others.
  The bank assesses perceived availability of helpful information or advice. The item bank does not use a time frame (e.g. over the past seven days) when assessing informational support. Informational Support instruments are available for adults (ages 18+)."
PROMIS Self-Efficacy at 2- and 6-weeks post randomization | 2- and 6-weeks post randomization
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy is described as the following according to HealthMeasures: "an individual's confidence in his/her ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. The PROMIS adult Self-Efficacy item banks assess self-reported current level of confidence in managing chronic conditions, including confidence in managing daily activities, managing emotions, managing medications and treatments, managing social interactions and managing symptoms. The self-efficacy item banks are universal rather than disease-specific. The respondent should be an adult (age 18+) and have at least one chronic health condition."
Generalized Anxiety Disorder 7-item (GAD 7) at 2- and 6-weeks post randomization | 2- and 6-weeks post randomization
  The Generalized Anxiety Disorder 7-item (GAD 7) is a seven item questionnaire, whereas a higher score is a higher indication of generalized anxiety disorder.
Post Traumatic Stress Disorder Checklist (PCL-5) at NICU discharge | at infant's NICU discharge, up to six (6) months.
  According to the National Center for PTSD, the Post Traumatic Stress Disorder Checklist (PCL-5) is described as the following: "The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including:
  * Monitoring symptom change during and after treatment
  * Screening individuals for PTSD
  * Making a provisional PTSD diagnosis The gold standard for diagnosing PTSD is a structured clinical interview such as the Clinician-Administered PTSD Scale (CAPS-5). When necessary, the PCL-5 can be scored to provide a provisional PTSD diagnosis."
NICU length of stay | from NICU admission to NICU discharge, up to six (6) months.
  Length of stay for the infant admitted to the Neonatal Intensive Care Unit (NICU) until they are discharged from the NICU.
Infant birth weight at NICU discharge | from NICU admission to NICU discharge, up to six (6) months.
  Weight of the infant admitted to the Neonatal Intensive Care Unit (NICU) at time of their NICU discharge.
App Usability and Satisfaction Scale at 2- and 6-weeks post randomization | 2- and 6-weeks post randomization
  A 5-point Likert scale and open-ended survey intended to analyze responses from those randomized to the intervention group.

OTHER OUTCOMES:
Clinically meaningful infant outcomes | From randomization through discharge, up to 6 months.
  Intraventricular hemorrhage (IVH), patent ductus arteriosus (PDA), sepsis, necrotizing enterocolitis (NEC), chronic lung disease (CLD)
Infant short-term outcomes | From randomization through discharge, up to 6 months.
  hearing test results
Infant short-term outcomes | From randomization through discharge, up to 6 months.
  length of stay
NICU Discharge Survey Results | Within 48 hours of NICU discharge, the survey will be completed.
  Results of the NICU Discharge Survey that were submitted by maternal participants. The survey contains questions about mode of infant feeding, and scaled and open-ended questions about their perception of communication and engagement with their health care team.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Osmundson, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will need to investigate feasibility